CLINICAL TRIAL: NCT00239486
Title: Evaluation of the Effect of Different Doses of Pramipexole on Subjective and Objective Symptoms of Idiopathic Restless Legs Syndrome (RLS).
Brief Title: Dose Finding Study of Pramipexole (Sifrol) in Patients With Idiopathic Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.515
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of different doses of pramipexole (Sifrol) on subjective and objective symptoms of idiopathic Restless Legs Syndrome (RLS) and also to determine the optimal dose of pramipexole in patients with RLS by polysomnography and evaluation of clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 18-80 years
2. Confident diagnosis of RLS according to International RLS Study Group criteria
3. RLS rating scale for severity score >15
4. PLM (during time in bed ) index at least 5 per hour
5. Weekly presence of RLS symptoms within last three months
6. Written Informed consent

Exclusion Criteria:

1. Women of childbearing potential, who do not use adequate protection such as barrier protection, intrauterine device, or hormonal (oral or subcutaneous) contraception
2. Postmenopausal women less than 6 months after last menses, surgically sterilised, oophorectomised or hysterectomised less than 3 months after operation and not using adequate protection
3. Women neither using adequate protection nor being postmenopausal and their partner is not sterilised at least 6 months post operation or does not use condom
4. Any women not having negative serum pregnancy test at screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109
Dates: Start 2002-10; Primary Completion 2004-04 (Actual); Study Completion 2004-04

PRIMARY OUTCOMES:
Reduction in periodic limb movements during time in bed index (PLMI) in the polysomnography (PSG). | 3 weeks

SECONDARY OUTCOMES:
Secondary outcomes of the study were other PSG-derived endpoints (changes in the RLS symptom rating scale (RLSRS), and patient reported outcomes). | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Finland Ky
Locations (1):
- NEURO, Helsinki, Finland